CLINICAL TRIAL: NCT02006108
Title: Non-invasive MR Imaging Diagnosis of Transplant Rejection
Brief Title: Imaging Kidney Transplant Rejection Using Ferumoxytol-Enhanced Magnetic Resonance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Lucile Packard Children's Hospital (Other)
Responsible Party: Principal Investigator, Heike E Daldrup-Link, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 94027
Record Dates: First submitted 2013-10-28; First posted 2013-12-09 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Renal Transplant Rejection
Keywords: kidney; transplant; rejection; Feraheme; ferumoxytol
MeSH Terms: conditions — Rejection, Psychology | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Feraheme (Experimental): Intravenous injection of Feraheme, 5 mg Fe/kg
  Interventions:
  Drug: Feraheme Procedure: MR Scan
  Interventions: Drug: Feraheme; Other: MRI-GE Healthcare 3 Tesla magnet

INTERVENTIONS:
Drug: Feraheme — Therapeutic classification: iron preparations. Use: Off-label use of ultrasmall paramagnetic iron nanoparticle as contrast agent for magnetic resonance imaging
  Other Names: Ferumoxytol
Other: MRI-GE Healthcare 3 Tesla magnet — All patients will undergo
  Other Names: Magnetic Resonance Imaging; MR Imaging

SUMMARY:
The goal of this study is to develop a non-invasive imaging test for in vivo detection of kidney transplant rejection. The hypotheses are that 1) Ferumoxytol-MRI can generate accurate estimates of tissue iron concentrations and tissue macrophages. 2) The signal given by a renal allograft on Ferumoxytol-MRI demonstrates significant differences between rejected and non-rejected transplants.

DETAILED DESCRIPTION:
In children with kidney transplants, immunologically mediated rejection is the major cause of allograft failure. Thus, the therapeutic success of kidney transplants is highly dependent on the ability to avoid rejection during both the acute and chronic phase after transplantation. Children with kidney transplants currently undergo at least three routine (protocol) biopsies during the first two years after the transplantation in addition to biopsies required to investigate deterioration of kidney function. These biopsies are invasive and nearly always require general anesthesia, causing anxiety and distress of the patients and their parents, as well as significant costs to our health care system. There is currently no non-invasive diagnostic tool capable of detecting rejection in vivo. Thus, the goal of this study is to develop a non-invasive imaging test for in vivo detection of kidney transplant rejection. The investigators propose to accomplish this goal by detecting macrophage infiltration in kidney transplants with iron oxide nanoparticle-enhanced MR imaging. Macrophages play a major role in transplant rejection. CD68-positive macrophages comprise approximately 50% of the infiltrating leukocyte population in renal allograft rejection, they co-localize with areas of tissue-damage and fibrosis, and are preponderant in more severe forms of rejection. The investigators hypothesize that iron oxide nanoparticle-enhanced MR imaging can detect differences in macrophage infiltrations in renal allografts undergoing rejection as opposed to allografts without significant rejection. This hypothesis is based on the bio-physical properties of intravenously injected superparamagnetic iron oxide nanoparticles, which are phagocytosed by tissue macrophages and cause strong signal effects on MR images.

The specific aims of the study are the following:

Aim #1. Technical Development of a Quantitative Susceptibility Mapping (QSM)-Sequence for in vivo MRI detection and quantification of iron oxide nanoparticle-labeled macrophages.This aim will focus on the technical development of Quantitative Susceptibility Mapping (QSM), a novel MR imaging pulse sequence that will be used to accurately quantify the tissue concentration of free ferumoxytol and ferumoxytol in macrophages in renal allografts. Based on pulse sequence optimizations of phantoms with known concentrations of free and cell-bound iron, we expect to generate accurate estimates of tissue iron concentrations and macrophages with the QSM-MRI method.

Aim #2. Detect rejection in kidney allografts with ferumoxytol-enhanced MRI. The investigators hypothesize that ferumoxytol can detect and quantify macrophages in kidney allografts, based upon the observation that iron oxide nanoparticles can be taken up by macrophages in malignant tumors. The investigators will evaluate the ability of ferumoxytol to map macrophage quantities in renal allografts, with histopathological correlation. We expect significantly higher ferumoxytol-MRI enhancement and macrophage quantities in rejected allografts compared to non-rejected allografts.

ELIGIBILITY:
Inclusion Criteria:

* Completed solid organ transplant with referral for transplant follow-up

Exclusion Criteria:

* Exclusion criteria comprise MR-incompatible metal implants, need of sedation (since an anesthesia is not supported by this), claustrophobia or hemosiderosis/hemochromatosis.

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heike E Daldrup-Link, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Feraheme: Intravenous injection of Feraheme, 5 mg Fe/kg
  Interventions:
  Drug: Feraheme Procedure: MR Scan
  Feraheme: Therapeutic classification: iron preparations. Use: Off-label use of ultrasmall paramagnetic iron nanoparticle as contrast agent for magnetic resonance imaging
  MRI-GE Healthcare 3 Tesla magnet: All patients will undergo
Period: Overall Study
Arm/Group | Feraheme
Started | 21
MR Imaging | 19
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Feraheme
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21
Number of Patients with Kidney Transplant [Count of Participants; unit: Participants] | 21
MRI Compatibility [Count of Participants; unit: Participants] | 21
Drug allergies, specifically against iron compounds [Count of Participants; unit: Participants] | 0
GFR [Mean (Standard Deviation); unit: ml/min/1.73 m2] — Population: overall study population is 21 patients we had 5 pts with rejection and 16 without. This is why the rows differ from overall
  ml/min/1.73 m2
    Rejection: number analyzed (Participants) | 5
    Rejection | 52 (24)
    Normal: number analyzed (Participants) | 16
    Normal | 90 (29)
Pregnancy [Count of Participants; unit: Participants] — Population: we checked all female participants for pregnancy and none was pregnant
  Participants
    number analyzed (Participants) | 9
    (all) | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiologically Detectable Differences in Signal Intensity Between Healthy and Rejected Kidneys, Measured Using T2* Maps
Description: According to the study hypothesis, macrophage infiltration into rejected kidneys will be significantly greater than in healthy kidneys; since macrophages are expected to phagocytose injected iron, there should be a detectable difference in signal intensity between healthy and rejected organs. This can be evaluated using semiquantitative T2* maps.
Time Frame: 24 hours to 7 days
Population: T2* value of transplant kidney
Measure: Mean (Standard Deviation); unit: ms (delayed postcontrast scans)
Arm/Group | Feraheme
Number analyzed (Participants) | 19
ms (delayed postcontrast scans)
  Rejection | 31.1 (14.4)
  No Rejection | 23.3 (5.4)

2. Secondary Outcome: Correlation of Cell-bound Iron Quantities on QSM Sequences With Macrophage and Iron Stains on Histopathology
Description: To evaluate our ability to quantify cell-bound iron using the novel QSM sequence, we use histopathological data showing 1) the iron content of renal tissue sampled, and 2) the level of macrophage infiltration of the renal tissue. We will perform iron and macrophage stains in biopsy tissues in order to determine this.
Time Frame: 3 weeks
Population: CD163 positive macrophages
Measure: Number; unit: correlation coefficient
Arm/Group | Feraheme
Number analyzed (Participants) | 19
correlation coefficient | 0

ADVERSE EVENTS:
Time Frame: Continuously for 30 minutes and on study completion.
Arm/Group | Feraheme
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT02006108/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02006108/SAP_001.pdf